CLINICAL TRIAL: NCT00716430
Title: Improving the Management of Non-ST Elevation Acute Coronary Syndrome: Systematic Evaluation of a Quality Improvement Programme
Brief Title: European Quality Improvement Programme for Acute Coronary Syndromes
Acronym: EQUIP-ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Uppsala University (Other); GlaxoSmithKline (Industry)
Responsible Party: Dr Marcus Flather, Royal Brompton Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EQUIP-ACS 1
Record Dates: First submitted 2008-07-11; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndromes; quality improvement
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- QI (Active Comparator): Quality Improvement Centres
  Interventions: Behavioral: Quality Improvement Programme
- Non-QI (No Intervention): No Quality Improvement Programme

INTERVENTIONS:
Behavioral: Quality Improvement Programme — Quality Improvement training programme
  Arms: QI

SUMMARY:
The main hypothesis to be tested is that the use of a quality improvement programme will lead to measurable improvements in the management of care and use of evidence based treatments for patients presenting to hospital with non-ST elevation acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

Patients with a good clinical history of ACS and at least one of the following:

* New or transient ST or T wave changes on the ECG consistent with acute myocardial ischaemia
* Elevation of troponin or other cardiac markers to levels indicative of myocardial necrosis according to local laboratory values

Exclusion Criteria:

* Evidence of persistent ST elevation on the ECG
* Use of early reperfusion therapy
* Patients >80 years
* Patients transferred from another hospital

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-12 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Composite of 7 outcome measures to assess aggregate potential for improvement in care using the QI programme:1:risk stratification within 24 hrs, 2:early coronary angiography, 3:anticoagulation, 4:beta-blockers, 5:statins, 6:ACE-inhibitors, 7:Clopidogrel | 10 months

SECONDARY OUTCOMES:
Clinical outcomes at discharge including death and myocardial infarction | 10 months
Estimated costs of care for patients | 10 months
Estimated costs and economic evaluation of potential cost-effectiveness of QI programme | 10 months

CONTACTS AND LOCATIONS:
Locations (37):
- France (8):
  - Centre Hospitalier de la region d'Annecy, Annecy
  - Centre Hospitalier de Chambery, Chambéry
  - Cardiology dept. B, CHU Hopital G. Montpied, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier de Riom Guy Thomas, Riom
  - Hopitaux Drome Nord de Romans-sur-Isere, Romans-sur-Isère
  - Centre Hospitalier d'Ussel, Ussel
  - Centre Hospitalier Pierre Bazin, Voiron
- Italy (5):
  - Ospedale M. Bufalini, Cesena
  - Ospedale Morgagni-Pierantoni, Forlì
  - Ospedale di Livorno, Livorno
  - Ospedale Generale Provinciale di Macerata, Macerata
  - Ospedale Civile di Mirano, Mirano
- Poland (10):
  - Szpital w Ciechanowie, Ciechanów
  - Szpital Zachodni, Grodzisk Mazowiecki
  - Szpital w Grojcu, Grójec
  - Swietofrzyskie Centrum Chorob Serca, Kielce
  - Szpital w Plocku, Płock
  - Radomski Szpital Specjalistyczny, Radom
  - Szpital Specjalistyczny SPZOZ w Radom, Radom
  - Szpital w Siedlcach, Siedlce
  - SP CSK- Medical University of Warsaw, Warsaw
  - Szpital we Wloclawku, Włocławek
- Spain (7):
  - Hospital Universitario Germans Trias, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Josep Trueta, Girona
  - Hospital Universitario Joan XXIII, Tarragona
  - Hospital de Terrassa, Terrassa-Barcelona
  - Hospital de Tortosa Virgen de la Cinta, Tortosa
- United Kingdom (7):
  - Antrim Area Hospital, Antrim
  - Barnet General Hospital, Barnet
  - Basildon Hospital, Essex
  - Warwick Hospital, Warwick
  - Royal Albert Edward Infirmary, Wigan
  - Yeovil District Hospital, Yeovil
  - York District Hospital, York

REFERENCES:
- [Derived] Flather MD, Babalis D, Booth J, Bardaji A, Machecourt J, Opolski G, Ottani F, Bueno H, Banya W, Brady AR, Bojestig M, Lindahl B. Cluster-randomized trial to evaluate the effects of a quality improvement program on management of non-ST-elevation acute coronary syndromes: The European Quality Improvement Programme for Acute Coronary Syndromes (EQUIP-ACS). Am Heart J. 2011 Oct;162(4):700-707.e1. doi: 10.1016/j.ahj.2011.07.027. PMID 21982663
- [Derived] Flather MD, Booth J, Babalis D, Bueno H, Steg PG, Opolski G, Ottani F, Machecourt J, Bardaji A, Bojestig M, Brady AR, Lindahl B. Improving the management of non-ST elevation acute coronary syndromes: systematic evaluation of a quality improvement programme European QUality Improvement Programme for Acute Coronary Syndrome: the EQUIP-ACS project protocol and design. Trials. 2010 Jan 14;11:5. doi: 10.1186/1745-6215-11-5. PMID 20074348